CLINICAL TRIAL: NCT04238130
Title: Evaluation Perioperative Dynamic Changes in ctDNA From Patients of Non-Small-Cell Lung Cancer Following Resection for Relapse Prediction
Brief Title: Evaluation ctDNA in Patients of Non-Small-Cell Lung Cancer Following Resection
Acronym: EVOLUTION
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hangzhou Repugene Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Other Study IDs: GASTO1058
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer (NSCLC); Resectable; Dynamic Monitoring; PEAC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Tissue, Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perioperative ctDNA Dynamic Monitoring Group: Samples were obtained at multiple pre-specified time points including before surgery (plasma samples)，during surgery after tumor resection (tumor samples) and after surgery(plasma samples were obtained every 6 months from ctDNA positive patients at baseline in the following 2 years)
  Interventions: Diagnostic Test: Perioperative ctDNA Dynamic Monitoring

INTERVENTIONS:
Diagnostic Test: Perioperative ctDNA Dynamic Monitoring — To apply ctDNA dynamic monitoring in early stage NSCLC patients with driver mutations positive at baseline

SUMMARY:
Circulating tumor DNA (ctDNA) is a promising biomarker for noninvasive assessment of cancer burden. In this study, PEAC (Personalized Analysis of Cancer) technology was performed to detect the driver gene mutations from plasma samples and matched tumor tissue samples were detected by NGS platform at baseline. Investigators also applied ctDNA dynamic monitoring using PEAC technology in early stage NSCLC patients with driver mutations positive at baseline, to evaluate the feasibility and their potential clinical application.

DETAILED DESCRIPTION:
Circulating tumor DNA (ctDNA) is a promising biomarker for noninvasive assessment of cancer burden. Advances in DNA sequencing technologies and our understanding of the molecular biology of tumours have resulted in increased interest in exploiting ctDNA as a tool to facilitate earlier detection of cancer and thereby improve therapeutic outcomes by enabling early intervention. In this study, PEAC (Personalized Analysis of Cancer) technology was performed to detect the driver gene mutations from plasma samples and matched tumor tissue samples were detected by NGS platform at baseline. Investigators aim to evaluate whether driver gene mutations detected by PEAC can replace tissue testing results in patients with stage I to Ⅲ NSCLC. Investigators also applied ctDNA dynamic monitoring using PEAC technology in early stage NSCLC patients with driver mutations positive at baseline, to evaluate the feasibility and their potential clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative histopathological diagnosis of TNM stage I to III NSCLC with R0 resection;
* No adjuvant chemotherapy, radiotherapy, targeted drug therapy or biotherapy after surgery;
* Men or women of age ≥18 years and <75 years old;
* Eastern Cooperative Oncology Group (ECOG) behavior status score 0 to 1.

Exclusion Criteria:

* Patients with other cancers other than NSCLC within five years prior to this study;
* Who can not get enough tumor histological specimens (non-cytological) for analysis;
* Human immunodeficiency virus (HIV) infection;
* NSCLC mixed with patients with small cell lung cancer;
* Pregnant or lactating women;
* There is a clear history of neurological or mental disorders, including epilepsy or dementia;
* Conditions that investigators think is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I to III Non-Small Cell Lung Cancer (NSCLC) with R0 resection
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Concordance between genomic alterations assessed by next-generation sequencing in tumor tissue and PEAC technology in circulating tumor DNA | 2 years after the last patient enrolled
  PEAC (Personalized Analysis of Cancer) technology was performed to detect the driver gene mutations from plasma samples and matched tumor tissue samples were detected by NGS platform at baseline.
ctDNA dynamic monitoring | 2 years after the last patient enrolled
  PEAC technology was performed to apply ctDNA dynamic monitoring in early stage NSCLC patients with driver mutations positive at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Si-Yu Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China